CLINICAL TRIAL: NCT00345514
Title: The Provider and Organization in Asthma Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michelle Cloutier, Professor of Pediatrics, UConn Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R01HL070785 (NIH); CCMC 01-111
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: Children; Self-efficacy; Organization; Process of care
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention)
- 2 (Active Comparator)
  Interventions: Behavioral: Behavioral Intervention Arm
- 3 (Active Comparator)
  Interventions: Behavioral: Organizational Interventions Arm

INTERVENTIONS:
Behavioral: Behavioral Intervention Arm — The arm emphasized individual provider behavior (interactive CME, feedback at the provider, clinic and program levels, expert modeling, academic detailing and opinion leaders)
  Other Names: Provider Intervention Arm
  Arms: 2
Behavioral: Organizational Interventions Arm — Leadership, team building, benchmarking at the clinic and program level
  Other Names: Organizational Arm
  Arms: 3

SUMMARY:
The purpose of this study is to examine the interaction between the personal attributes of clinicians and the organizations in which they work and the effect of interventions on their ability to implement an asthma disease management program. +

DETAILED DESCRIPTION:
Less than 20% of primary care providers adhere to national asthma guidelines. Interventions to improve provider adherence to guidelines have had modest success. We believe that changing provider behavior must be viewed in the context of the provider's environment. We hypothesize that providers who are most successful in implementing and sustaining asthma management programs will have a set of personal attributes, related to asthma, characterized by readiness to change, high self-efficacy, positive outcome expectancies and high outcome value AND will work within organizations that facilitate and support such activities. We propose a two phase study. In Phase 1 (Year 1) survey instrument development and testing and provider meetings to discuss the interventions will occur. Providers in 49 practices/clinics that are using an asthma management program called Easy Breathing, will complete these surveys that will characterize the organization and organizational culture of the clinics/practices and the provider personal attributes surrounding asthma. In Years 2-5, a randomized, controlled study of either a behavioral intervention, an organizational intervention or no intervention (control) will be performed in 36 of these clinics/practices. Clinics/practices in the behavioral arm will receive an intervention consisting of expert modeling, program-, clinic- and provider-specific feedback, and use of opinion leaders and academic detailing. Clinics/practices in the organizational arm will receive an intervention consisting of benchmarking, leadership capability training and team building and incentives/ rewards. The primary outcome variable is the number of Easy Breathing surveys completed by provider and by clinic/unit of time. We have previously shown that enrollment in Easy Breathing (which was adapted directly from the national asthma guidelines) as demonstrated by completion of a survey is a surrogate indicator of inhaled corticosteroid use and is associated with decreased medical services utilization. This study will thus investigate the complex interactions between provider personal attributes and the organization and the effect of targeted interventions on provider performance to implement an asthma disease management program. These data will then be used in future studies to determine how to better tailor interventions in a cost constrained environment.

ELIGIBILITY:
Inclusion Criteria:

* Must have used Easy Breathing Disease Management Program for more than one year.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Number of Easy Breathing Surveys Distributed | 4 years

SECONDARY OUTCOMES:
Organizational Culture | baseline; 12 months and 36 months after intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Cloutier, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States